CLINICAL TRIAL: NCT07269119
Title: Designing Deaf-MET: A Deaf-Accessible Pre-Treatment for Alcohol Use Disorder
Brief Title: Piloting a Deaf Accessible Pre-Treatment for AUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Alexander Wilkins, Assistant Professor, Dept of Psychiatry and Behavioral Sciences, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002259; K23AA029466 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; deaf
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm: Deaf-MET Intervention (Experimental): Participants in the experimental arm will receive Deaf-MET, a culturally and linguistically accessible adaptation of Motivational Enhancement Therapy (MET) for Deaf adults with high-risk alcohol use. MET is a client-centered counseling approach that enhances motivation for change by exploring and resolving ambivalence, using reflective listening, feedback, and collaborative goal-setting. Deaf-MET will be delivered in American Sign Language and incorporates visual handouts, plain language materials, and filmed educational content adapted from the original MET protocol into ASL teaching stories. Sessions are offered in-person or via telehealth.
  Interventions: Behavioral: Deaf-MET

INTERVENTIONS:
Behavioral: Deaf-MET — Deaf-MET is a culturally and linguistically accessible adaptation of Motivational Enhancement Therapy (MET) for Deaf adults with high-risk alcohol use

SUMMARY:
This pilot study will evaluate the feasibility, acceptability, and preliminary efficacy of an adaptation of Motivational Enhancement Therapy (MET) titled "DeafMET", intended for Deaf adults with high-risk alcohol use. In this single intervention cycle, 10 Deaf participants will receive the DeafMET intervention delivered either in-person or via telehealth. Primary outcomes include change in participants' stage of change regarding alcohol use and measures of recruitment, retention, satisfaction, and adherence. Findings will inform further refinement of the intervention and planning for future research.

DETAILED DESCRIPTION:
This study will conduct the first clinical pilot of DeafMET, a Deaf-accessible adaptation of Motivational Enhancement Therapy (MET) for alcohol use disorder (AUD) in Deaf adults. The U.S. Deaf community-over one million Americans who use American Sign Language (ASL)-experiences disproportionate rates of high-risk alcohol use and barriers to behavioral health care. Studies indicate that Deaf adults face significantly higher rates of lifetime problem drinking and are less likely to access evidence-based AUD treatment compared to their hearing peers. Unique challenges, such as limited English literacy, lack of available mental health resources in ASL, and low health literacy, contribute to poor health outcomes and marginalization within existing care systems.

While motivational interviewing and enhancement therapies are widely validated for treating substance use disorders in hearing populations, there are currently no evidence-based behavioral health interventions specifically adapted for Deaf individuals. Existing AUD treatments rely heavily on written English materials and verbal processing, limiting their accessibility and effectiveness among ASL users. Research demonstrates that Deaf people's average English reading level is at grade four, and health-related comprehension closely matches that of non-English-speaking immigrants. These disparities underscore the urgent need for linguistically and culturally tailored treatment protocols.

To address these barriers, the study team developed and refined the DeafMET prototype through comprehensive literature review, stakeholder input, and community engagement. The intervention features:

* Deaf-friendly client materials such as visual handouts revised for plain text and created with input from Deaf artists
* Translated ASL educational content
* Interactive components leveraging visual and narrative strategies that are accessible to Deaf clients with varied health literacy

The adaptation was developed in collaboration with Deaf clinicians, persons in recovery, and other stakeholders to maximize relevance, clarity, and engagement. The study design is a single-cycle pilot enrolling 30 Deaf adults who report past-month high-risk alcohol consumption and related problems. Recruitment will utilize networks within Deaf-serving organizations, behavioral health programs, and community outreach to ensure broad reach. Participants will receive the DeafMET intervention delivered by a Deaf therapist fluent in ASL. Sessions may be conducted in-person or remotely.

After meeting with the PI to determine study eligibility and provide informed consent, participants will complete the pre-intervention assessments. The participant will be sent a link to REDCap where they will complete a one-time demographic survey and 9 measures, estimated to take 1.5-2 hours. These measures have been translated into American Sign Language and participants will have access to both the ASL and written English versions of each measure.

Following completion of the pre-intervention measures, the DeafMET intervention will be administered either in-person or via Zoom. In-person sessions will be held in a private room in UMass Chan's Chang Building on the Shrewsbury campus. Choice of in-person or virtual sessions will depend on the potential participants' preference, location of residence, and transportation needs. Ideally, participants will be balanced across session format. In-person sessions will be conducted at the Chang Building on UMass' Shrewsbury campus in a private room designed for research purposes. Virtual sessions will be held either in the PI's office in the Chang Building or in another private room. There will be six sessions, each running for 1 hour, occurring on a biweekly basis. Participation in this trial is expected to last 13 weeks, inclusive of pre-intervention assessment and exit interview. Participants will be provided with an adapted psychotherapy intervention at no cost. The original intervention, MET, has been used successfully in both research and clinical settings with various populations since its inception in the 1990s. Adaptations were made to both the session structure and order as well as materials to better align with the needs of the deaf community. In addition, both the original MET and the current adaptation are designed to be brief interventions to be administered prior to other types of more intensive therapies or treatments, in order to boost internal motivation in recovery from AUD. If participants are interested in immediately starting long-term we will recommend they not participate in the study and instead provide resources to find local therapists who take their insurance. We can also provide the option to participate in the study while providing resources to start seeing a local therapist after they finish study participation.

All sessions will be recorded for consistency of session format. However, only 25% of each participant's sessions will be reviewed. The sessions will be reviewed for PI's fidelity to motivational interviewing principles using the Motivational Interviewing Competency Assessment (MICA) system. The research coordinator will receive training on the MICA coding system via the Motivational Interviewing Network of Trainers.

The first session will be the introductory session. The purpose of this session is to establish rapport, set the schema of MET and our work together, allow the client to share their reasons for coming and past experiences with therapy and/or recovery.

The 2nd session will be where the value card sort activity is completed. The purpose of this session is to complete the value card activity with the clients and answer any follow up questions from the first session. The focus of this session is to increase client's sense of empowerment and understanding of where they stand in life and start them thinking about the role alcohol plays in their life.

The 3rd and 4th sessions will be the assessment/interview sessions. The purpose of these sessions is to administer all of the assessments and interview questions that will be used to complete the personal feedback report.

In between the 3rd and 4th sessions, the participant will complete the mid-intervention assessments. They will again be sent a link to REDCap where they will complete the same 9 measures as the pre-intervention assessment.

The 5th session is where the personal feedback report will be reviewed. The purpose of this session is to review progress, share the Personal Feedback Report (PFR) based on prior assessments, and begin transitioning into Phase 2 of MET: strengthening commitment to change. If the client is interested, a partner or support person may join to provide their perspective and support.

The 6th and final session is to deepen the conversation. This session serves to deepen exploration of motivation, especially if the client is still ambivalent or has not yet committed to change. It offers space to continue reflecting on feedback, life goals, and the role of alcohol. For clients already engaging in change, the session can support ongoing commitment and planning.

After completing the 6th session, the participant will again be sent a link to REDCap where they will complete the same 9 measures as the pre- and mid-intervention assessment. In addition, the research coordinator will complete a semi-structured qualitative interview with each participant to elicit their feedback on all parts of the DeafMET intervention.

ELIGIBILITY:
Inclusion Criteria:

* self-identification as a Deaf ASL user
* age 18+
* ability to access Zoom for screening, intervention delivery, and repeated assessment procedures
* problematic alcohol consumption, drinking behaviors, and alcohol-related problems" as identified by the AUD Identification Test (AUDIT), past-month referent time period: score at least 8 for men or at least 6 for women

Exclusion Criteria:

* Incapacity to consent due to guardianship or conservatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
University of Rhode Island Change Assessment | From enrollment to end of participation at 3 months
  URICA measures a patient's readiness to change using a self-reported questionnaire that categorizes the patient into one of the 4 following stages: precontemplation, contemplation, action, or maintenance. Potential scores range from -2 to 14. Scores below 8 indicate precontemplation. Scores between 8-11 indicate contemplation. Scores above 11 indicate preparation or action stage.
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES 8A) | From enrollment to end of treatment at 3 months
  The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) is an instrument designed to assess motivation for change in problem drinkers. There are three scales: Recognition (score range 7-35), Ambivalence (score range 4-20), and Taking Steps (score range 8-40). For all scales, a higher score is better in that they 1) recognize they have a drinking problem, 2) are thinking about their drinking's effect on people, and 3) are actively taking steps to change.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test | From enrollment to end of treatment at 3 months
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Possible scores range from 0-40, with a 0 indicating no alcohol consumption, 1-7 indicating low risk alcohol consumption, 8-14 indicating higher risk alcohol consumption, and above 15 indicating the likelihood of at least moderate alcohol use disorder.
Alcohol Timeline Followback | From enrollment to end of treatment at 3 months
  The Timeline Follow Back is a calendar that allows a clinician to get an estimate of an individual's daily drinking habits over a given time period. There is no scoring scale for this measure, it is simply used to count the number of days someone drank over the last month as well as how many drinks they had.
Comprehensive Effects of Alcohol- Brief | From enrollment to end of treatment at 3 months
  The Brief Comprehensive Effects of Alcohol questionnaire (B-CEOA) is a 15-item assessment of expectancies concerning alcohol effects. Respondents indicate their degree of agreement that a particular effect will likely occur if they drink, using a 1-4 scale (1 = disagree, 4 = agree). Scores range from 15-60, with higher scores indicating experiencing more negative effects from drinking alcohol.
Penn Alcohol Craving Scale | From enrollment to end of treatment at 3 months
  The Penn Alcohol Craving Scale (PACS) is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week. Scores range from 0-30, with a higher score indicating a stronger craving to drink alcohol.
California Psychotherapy Alliance Scale | From enrollment to end of treatment at 3 months
  The California Psychotherapy Alliance Scale (CALPAS) is a self-report measure of therapeutic alliance. The CALPAS includes items tapping the client's commitment to therapy, his or her capacity to undertake work, the therapist's understanding/involvement in therapy, and the dyad's agreement on goals/strategies. These items attempt to capture the nature of the interaction between the therapist and client, which is central in the concept of the alliance. Scores range from 12 to 84 with a higher score indicating a stronger therapeutic allicance.
Social Support Questionnaire- 6 | From enrollment to end of treatment at 3 months
  The Social Support Questionnaire 6 (SSQ6) is a brief self-report measure of perceived social support. It consists of 6 questions that ask respondents to list up to 9 people who provide them with different types of support and rate their satisfaction with the overall support received. The questionnaire provides a measure of perceived social support availability (number of supporters listed) and satisfaction with available support. Scores are calculated for number of supporters, satisfaction, and number of family supporters to assess an individual's social support network. Higher scores indicate a better social support network.
Change talk assessment | From enrollment to end of treatment at 3 months
  The Motivational Interviewing Competency Assessment (MICA) is used to see how well a clinician uses motivational interviewing (MI) techniques during sessions about health behavior change or treatment. It is scored by reviewing a conversation (at least 8 minutes) between the clinician and one client. MICA focuses on skills like working in partnership, encouraging change, showing empathy, and supporting the client's choices. Trained reviewers rate how often and how well the clinician uses these skills. Scores show overall MI competency. The results help clinicians improve their ability to use MI in practice. There are seven categories (scores range from 1-5) and one composite score (scores range from 2-12) where higher scores indicate better fidelity to MI principles.

OTHER OUTCOMES:
Client Exit Interview | Upon completion of treatment at 13 weeks
  An optional exit interview will be conducted with each participant to elicit thoughts and feedback on the DeafMET intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wilkins, PhD, MSCI, Principal Investigator — UMass Chan Medical School

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit and share data with the NIAAA Data Archive, a data repository housed within the National Institute on Mental Health (NIMH) Data Archive (NDA), per the requirements set forth in NOT-AA-23-002 (grants.nih.gov/grants/guide/notice-files/NOT-AA-23-002.html). All data will be de-identified before submission to the data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The investigators will submit data on or before the NDA submission due dates (April 1 and October 1 each year) in accordance with the applicable Data Sharing Terms and Conditions of award.
Access Criteria: Can be accessed via the NIAAA Data Archive (NIAAADA)
URL: https://nda.nih.gov/niaaa